CLINICAL TRIAL: NCT00714233
Title: Treatment of Polycystic Ovary Syndrome (POS) in Overweight Adolescents
Brief Title: Treatment of Adolescent Polycystic Ovary Syndrome (PCOS)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Rochester (Other)
Responsible Party: Principal Investigator, Kathleen M. Hoeger, MD, Professor, University of Rochester
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: RSRB # 09354
Record Dates: First submitted 2008-07-08; First posted 2008-07-14 (Estimated); Results first posted 2011-09-16 (Estimated); Last update posted 2015-05-15 (Estimated); Status verified 2011-05

CONDITIONS: Polycystic Ovary Syndrome
Keywords: Polycystic Ovary Syndrome; Overweight Adolescent Girls; Irregular Menstrual Cycles
MeSH Terms: conditions — Polycystic Ovary Syndrome; Menstruation Disturbances | interventions — Metformin; drospirenone and ethinyl estradiol combination

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Experimental): Metformin
  Interventions: Drug: Metformin
- 2 (Experimental): Oral Contraceptive Pills
  Interventions: Drug: Oral Contraceptive Pills (Yasmin)
- 3 (Active Comparator): lifestyle modification program
  Interventions: Behavioral: Lifestyle Modification
- 4 (Placebo Comparator): placebo to active metformin arm
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Metformin — Metformin 425mg. capsules, 2 capsules BID x 24 weeks
  Arms: 1
Drug: Oral Contraceptive Pills (Yasmin) — Yasmin oral contraceptive tabs; 1 tab daily x 24 weeks
  Other Names: Yasmin oral COntraceptive tabs
  Arms: 2
Behavioral: Lifestyle Modification — weekly classes x 24 weeks for training in diet, exercise and behavior modification skills
  Arms: 3
Drug: placebo — placebo to the active metformin arm. 2 capsules BID x 24 weeks.
  Other Names: pharmacy matched placebo capsules
  Arms: 4

SUMMARY:
A 24 week study to compare the use of Metformin, birth control pills and a carefully planned intensive lifestyle program that includes weight loss and exercise. These approaches will be compared to placebo (a pill that contains no active substances. Metformin, birth control pills and the lifestyle management program will be used on this research study to compare their ability to:

1. reduce fasting glucose levels
2. reduce androgen hormone levels
3. improve sex steroid binding, and
4. improve lipids (fatty substances in the blood)

DETAILED DESCRIPTION:
Polycystic ovary syndrome (PCOS) is a condition associated with irregular menstrual cycles, (due to lack of regular ovulation), and evidence of elevated androgen (male hormone) levels, such as unwanted hair growth or acne. This condition often becomes recognized at the time of puberty. The standard treatment for this condition is oral contraceptive pills, which are used not for contraception, but to cause a regular, monthly bleeding pattern.

Many adolescents with PCOS have increased levels of insulin, a hormone that controls the body's sugar balance. These increased insulin levels may play a role in the development of polycystic ovary syndrome. There are several medications now available, which can decrease the insulin levels by improving the action of insulin in the body. Metformin is one of these drugs. Metformin is a drug currently used in the management of diabetes to control blood sugar. It is hoped that by lowering the insulin levels some of the symptoms of polycystic ovary syndrome, such as the lack of regular periods and unwanted hair growth, can be reversed or diminished.

ELIGIBILITY:
Inclusion Criteria:

* Menstrual irregularity defined as cycle length > 45 days
* Overweight as BMI > 25
* Clinical evidence of hirsuitism or acne
* Testosterone > 50ng/dL

Exclusion Criteria:

* History of diabetes mellitus
* History of Cushing's disease
* History of hyperprolactinemia
* Untreated hypo or hyperthyroidism
* History of adrenal hyperplasia
* Significant renal impairment
* Received oral contraceptives, estrogen or progestin or other drugs known to effect lipoprotein metabolism within 2 months of starting the study
* Exercise > 10 hours per week

Ages: 12 Years to 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 43 (Actual)
Dates: Start 2002-08; Primary Completion 2004-04 (Actual); Study Completion 2007-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen M Hoeger, MD, Principal Investigator — University of Rochester

RESULTS

PARTICIPANT FLOW:
Groups:
- Metformin: Randomized to Metformin 1700mg daily for 24 weeks
- Oral Contraceptive: Randomized to Oral Contraceptive Pills for 24 weeks. Monitored monthly for compliance
- Lifestyle Counseling: lifestyle modification program consisting of nutritional counseling and dietary counseling meeting weekly
- Placebo to Metformin: randomized to placebo pill identical to active metformin arm
Period: Overall Study
Arm/Group | Metformin | Oral Contraceptive | Lifestyle Counseling | Placebo to Metformin
Started | 10 | 11 | 11 | 10
Completed | 6 | 10 | 10 | 6
Not Completed | 4 | 1 | 1 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Metformin | Oral Contraceptive | Lifestyle Counseling | Placebo to Metformin | Total
Number analyzed (Participants) | 10 | 11 | 11 | 10 | 42
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 10 | 11 | 11 | 10 | 42
  Between 18 and 65 years | 0 | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 16 (1.7) | 15.4 (1.4) | 15.4 (1.2) | 15.4 (1.7) | 15.6 (1.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 11 | 11 | 10 | 42
  Male | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 10 | 11 | 11 | 10 | 42

OUTCOME MEASURES:

1. Primary Outcome: Measure Number of Adolescent Girls With PCOS Who Can be Successfully Recruited Into a Randomized Clinical Trial That Includes Lifestyle Modification
Description: The measure is to determine a number of successfully recruited overweight or obese adolescents to a randomized trial of lifestyle therapy in the community of Rochester, NY
Time Frame: 24 week
Population: Analysis was a description of number of recruited subjects.
Measure: Number; unit: participants
Arm/Group | Metformin | Oral Contraceptive | Lifestyle Counseling | Placebo to Metformin
Number analyzed (Participants) | 10 | 11 | 11 | 10
participants | 10 | 11 | 11 | 10

2. Secondary Outcome: Weight Loss in Lifestyle Intervention Group
Description: In the adolescent women assigned to the lifestyle program, did the intervention program obtain weight reduction as measured by change in BMI
Time Frame: baseline and 24 weeks
Population: Analysis per protocol
Measure: Mean (Standard Deviation); unit: kg/m^2
Groups:
- Lifestyle Program: Subjects enrolled in a nutrition and exercise program
Arm/Group | Lifestyle Program
Number analyzed (Participants) | 8
kg/m^2 | -1.1 (6.6)
Statistical Analysis 1: Comparison: Lifestyle Program; Paired t-test to analyze BMI at baseline and 24 weeks; Test type: Superiority or Other; p < 0.05, t-test, 2 sided

3. Secondary Outcome: Change in Free Androgen Index (FAI)
Description: Secondary measures of reduction in androgen measures of the different treatment arms. This is a ratio of total testosterone to sex hormone binding globulin (SHBG). The lower values correlate with lower amount of free testosterone. FAI <4 is consistent with a normal range.
Time Frame: baseline and 24 weeks
Population: analysis per protocol
Measure: Mean (Standard Deviation); unit: total T/SHBG
Groups:
- Metformin: Group assigned to metformin with free androgen index measured
- Oral Contraceptive: group assigned to oral contraceptive for 24 weeks
- Lifestle: Those assigned to a nutrition and exercise program
- Placebo to Metformin: Matched to metformin pill
Arm/Group | Metformin | Oral Contraceptive | Lifestle | Placebo to Metformin
Number analyzed (Participants) | 6 | 10 | 8 | 10
total T/SHBG | -0.1 (3.2) | -16.7 (8) | -13.7 (10.9) | 1.2 (12.3)

4. Secondary Outcome: Change in SHBG
Description: Measurement of SHBG by treatment group pre and post intervention
Time Frame: baseline and 24 weeks
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Metformin | Oral Contraceptive | Lifestyle Counseling | Placebo to Metformin
Number analyzed (Participants) | 6 | 10 | 8 | 10
ratio | 2.6 (8.6) | 77 (38.4) | 17.6 (18.3) | 2 (8.4)

5. Secondary Outcome: Triglyceride Concentration by Treatment Group
Description: Change in triglyceride measures pre and post intervention as representative of lipid changes by treatment group; metformin, lifestyle intervention, oral contraceptive or placebo
Time Frame: baseline and 24 weeks
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Metformin | Oral Contraceptive | Lifestyle Counseling | Placebo to Metformin
Number analyzed (Participants) | 6 | 10 | 8 | 10
mg/dL | -22.3 (24.1) | 4.6 (41) | 2.2 (36.4) | -6.6 (27.8)

6. Secondary Outcome: Change in Fasting Glucose
Description: Change in fasting glucose concentration by treatment group pre to post intervention
Time Frame: baseline and 24 weeks
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Metformin | Oral Contraceptive | Lifestyle Counseling | Placebo to Metformin
Number analyzed (Participants) | 6 | 10 | 8 | 10
mg/dL | -6.7 (10.3) | 6.9 (8.7) | 0.4 (7.2) | -1.1 (7.2)

ADVERSE EVENTS:
Arm/Group | Metformin | Oral Contraceptive | Lifestyle Counseling | Placebo to Metformin
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/11 | 0/11 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/11 | 0/11 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No